CLINICAL TRIAL: NCT00207259
Title: Study of Complementary Therapies in Men Receiving Radiation Therapy for Prostate Cancer: A Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Clair Beard, Attending Physician, Vice-Chair, Genitourinary Radiaton Oncology, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-005
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Reiki; Relaxation Response; Cognitive Restructuring; Feasibility
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutic Touch; Cognitive Restructuring; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Standard weekly treatments with radiation oncologist and nurse. All control patients offered intervention at end of 8-week course of radiotherapy.
- Relaxation Therapy (Experimental): Weekly relaxation therapy with PhD psychologist and home cognitive restructering practice
  Interventions: Behavioral: Reiki & Relaxation Response Therapy with Cognitive Restructuring
- Reiki (Experimental): Weekly Reiki therapy with a Reiki therapist, involves laying of the therapist's hands on the patient to rechannel energy, considered pleasant and calming
  Interventions: Behavioral: Reiki & Relaxation Response Therapy with Cognitive Restructuring

INTERVENTIONS:
Behavioral: Reiki & Relaxation Response Therapy with Cognitive Restructuring — Relaxation Therapy: Practice of focus on breathing or repeated word while ignoring random thoughts without bias. Designed to lower heart rate, blood pressure and stress.
  Reiki: Practice of laying on hands by a Reiki therapist in order to channel patient's energy, considered calming and pleasant.
  Other Names: Relaxation Therapy; Reiki therapy
  Arms: Reiki; Relaxation Therapy

SUMMARY:
Randomized clinical study of two CAM therapies, 1) Reiki and 2) Relaxation Response Therapy with Cognitive Restructuring counseling (RRT with CR), compared to an education-only control arm in patients about to begin an eight-week course of external beam radiotherapy (EBRx) for prostate cancer.

Generally, we would like to examine the feasibility of studying Reiki and RRT with CR in patients with prostate cancer, and to obtain preliminary results on the effectiveness of these treatments compared to controls.

Specific objectives:

1. Determine the proportion of eligible patients who agree to participate in the study
2. Measure compliance with CAM therapy interventions
3. Measure compliance with physiologic and psychological outcome measurement assessments
4. Assess differences between experimental and control groups on measures on depression, anxiety, quality of life, salivary cortisol levels and an immunomarkers

DETAILED DESCRIPTION:
Part of the mission of the Dana-Farber/Brigham and Women's Cancer Center is to enhance the quality of life for cancer patients and their families. Treatments and therapies specifically designed to address changes in the cognitive, emotional and spiritual realm experienced by patients as they attempt to cope with cancer are now routinely offered in addition to standard and experimental medical therapies and fall into the realm of complementary and alternative medicine (CAM) and support. Our patients may participate in support groups; work with a social worker, psychologist or psychiatrist privately; learn about diet in seminars or meet with a dietician; participate in art or music therapy; or participate in the many programs offered by the Leonard P. Zakim Center, which include Reiki therapy, acupuncture, acupressure, massage and therapeutic touch. All of these services are provided with the hope that the participants derive some benefit, however intangible. That cancer patients experience significant short- and long-term psychological distress associated with their cancer diagnosis and treatment is well documented.1-4 Most feel a strong sense of lost self-control and experience disturbances in appetite, sleep, concentration, and stamina.5-9 Anxiety and depression appear to be almost ubiquitous with a cancer diagnosis, including those men diagnosed with prostate cancer.8,10-12 This may explain the prevalence of prostate cancer support groups, internet sites and self-help books. However, we have little precise information on our own prostate cancer population with regards to the choices they make regarding CAM and no information on how CAM therapies affect them.

There are some data on the use of CAM in other prostate cancer populations.13-16 In a study of 1,099 men, the prostate cancer diagnosis prompted 23.5% of the sample to start using some form of CAM for health, and 67% of the group reported having used some form of CAM for prostate health before being diagnosed.17 The study included 14 herbal or dietary therapies and 16 mind-body therapies. There were demographic differences between patients who opted for CAM use and those who did not. Patients choosing CAM were more likely to be white versus not, and more likely to be college-educated versus not. The latter variable was particularly significant in this analysis. A second study of patients living in and around San Francisco reported on 543 prostate cancer patients who completed a 30-minute telephone interview regarding complementary and alternative medicines.14 Overall, 30% of the participants used at least one type of complementary or alternative medicine. CAM users were younger than non-users and likely to be college graduates. In this group, herbal remedies and mental health approaches were the most commonly utilized, followed by dietary changes. Twelve percent of the population used two or more CAM approaches.11

For our own study, we chose to look at two forms of CAM, Reiki and relaxation response therapy (RRT). These two were chosen as we had some evidence of utilization within our own cancer population. Reiki treatment is given at the Zakim Center. In the four years since the Zakim Center opened, there have been approximately 300 patient visits for Reiki therapy. Reiki is an energy healing method discovered in the late 1800s in Japan. The word Reiki is made up of two Japanese words: Rei, an unlimited universal power of force that acts in all created matter; and Ki, a living spirit energy that applies to the physical principle of life. Licensed Reiki Masters perform Reiki. All of the Reiki Masters at the Zakim Center are also registered nurses. Subjects often express an enhanced sense of well-being and relaxation after a Reiki session, according to the Reiki practitioners, and most return for at least one more session. Led by Susan DeCristofaro, the Reiki experience at the Zakim Center has been standardized. Here, Reiki is given for acute and chronic pain, headache, depression, anxiety, nausea, vomiting and insomnia. The fee for a Reiki session is $55.00. However, the effects of receiving Reiki have not been subjected to rigorous scientific study. In a review of energy healing, eleven studies looking at Reiki were reviewed. Of these, seven showed a beneficial effect,18-22 three showed no effect21,23,24 and one had a negative effect.25 We believe, after review of this data, that there are many unanswered questions about this treatment.

The second CAM of interest to us was relaxation response therapy (RRT), described and pioneered at the Mind/Body Medical Institute, directed by Herbert Benson, MD. The Mind/Body Medical Institute is an independent, nonprofit organization dedicated to the study of mind/body interactions, including RRT. Three to four hundred cancer patients per year participate in programs at the Mind/Body Medical Institute. Interventions using RRT in combination with cognitive restructuring (CR) counseling are commonly employed and are felt to be 'successful' in cancer patients by the practitioners who deliver them.

The term "relaxation response" was first coined in 1974.26,27 This technique has two characteristics: repetition of a word or phrase and a disregard of everyday thoughts. The elicitation of the RR down-regulates the sympathetic nervous system. It is characterized by reductions in oxygen consumption, respiratory rate, blood pressure, heart rate and arterial blood lactate. The mind/body state achieved with RR is consistent with a wakeful, hypometabolic physiological state.28 EEG studies clearly differentiate the RR from sleep.29 PET30 and fMRI31 studies have correlated specific regional changes in brain activity with the elicitation of the RR. When the patient is in a relaxed state, the therapist focuses on helping him to identify emotions, negative thoughts or anxieties and assisting him to deal with these thoughts in a more constructive way. This is called "cognitive restructuring" and it is an integral part of RT.

RRT is believed to be a useful therapeutic intervention in numerous conditions including: headache;32-34 premature ventricular contractions in stable ischemic heart disease or hypertension;35-38 anxiety;39,40 stress symptoms;41 cardiac surgery;37 pain relief and anxiety reduction in femoral arteriography;42 premenstrual syndrome;43 infertility;44 psychosomatic complaints;45 chronic pain;46-48 and insomnia.29 Other investigators have also found that RRT techniques were effective in the treatment of rheumatoid arthritis. The fee for RT with cognitive restructuring is $100.00 per hour, paid for privately or through insurance.

Thus, we identified two reasonably mature CAM therapies offered and apparently utilized by our own patients, paid for by the patients and their insurance providers, believed by the practitioners to be beneficial to patients but without much solid evidence to support their use. We also know that prostate cancer patients have a high level of interest in CAM. With this in mind, we applied for and received a grant from the Advanced Medical Research Foundation and submitted a protocol to the Dana-Farber/ Harvard Cancer Center Internal Review Board with the primary aim of assessing the feasibility of recruiting and maintaining enrollment in CAM therapy during an 8-week course of RT and a 2-month follow-up period. Our protocol was accepted, #05-005, and is now accruing patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 30
2. Histologic documentation of prostate cancer (no time limit)
3. Gleason score assignment is mandatory prior to entry
4. ECOG Performance Status of 0, 1, or 2
5. Clinical Stage Tl - T4 adenocarcinoma of the prostate
6. Planned androgen suppression therapy prior to an eight-week course of external beam radiotherapy
7. Signed Informed Consent

Exclusion Criteria:

1. Prior pelvic radiotherapy
2. Evidence of metastatic disease
3. Currently receiving ongoing psychotherapy or antidepressive medications
4. Non-English speaking

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Obtain preliminary results on the effectiveness of these treatments compared to controls | Measurements taken at multiple time points
  QOL testing performed at four time points

CONTACTS AND LOCATIONS:
Overall Officials: Clair Beard, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States